CLINICAL TRIAL: NCT07354191
Title: Outcome of Multiple Myeloma Associated With Autoimmune Hemolytic Anemia: Cross-sectional Study
Brief Title: Outcome of Multiple Myeloma Associated With Autoimmune Hemolytic Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Hussein, Lecturer, New Valley University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MAIHA
Record Dates: First submitted 2025-11-21; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Coombs Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MM patients (Experimental): the prevalence of AIHA in MM patients and determine its impact on clinical presentation and outcome of the disease
  Interventions: Diagnostic Test: direct antiglobulin test (DAT); Diagnostic Test: Indirect antiglobulin test (IAT)

INTERVENTIONS:
Diagnostic Test: direct antiglobulin test (DAT) — Serum sample
Diagnostic Test: Indirect antiglobulin test (IAT) — Serum sample

SUMMARY:
Autoimmune hemolytic anemia (AIHA) is a highly heterogeneous disease due to increased destruction of autologous erythrocytes by autoantibodies with or without complement involvement. Other pathogenic mechanisms include hyper-activation of cellular immune effectors, cytokine dysregulation, and ineffective marrow compensation.

DETAILED DESCRIPTION:
AIHAs may be primary or associated with lymphoproliferative and autoimmune diseases, infections, immunodeficiencies, solid tumors, transplants, and drugs. The direct antiglobulin test is the cornerstone of diagnosis, allowing the distinction into warm forms (wAIHA), cold agglutinin disease (CAD), and other more rare forms. Multiple myeloma (MM), on the other hand, is characterized by a clonal expansion of plasma cells in bone marrow, causing bone tissue destruction, renal failure and hematopoietic suppression. Although the association of MM and anemia is common, AIHA as the anemic manifestation of MM is rare. This prospective study will be conducted to detect the presence of AIHA in MM patients and its impact on clinical presentation and outcome of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of multiple myeloma

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Measure prevalence of AIHA in MM patients . | baseline
  Number of MM patients with AIHA
Detect impact on International Prognostic Scoring System | baseline
  relation of the presence of AIHA to the scoring system of the patient
Detect impact on outcome | through study completion, an average of 1 year
  Number of patient with AIHA regarding in each response group CR, PR, PD

SECONDARY OUTCOMES:
Identify complications of AIHA IN MM | through study completion, an average of 1 year
  number pf complications related to AIHA in each patien

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barcellini W, Zaninoni A, Giannotta JA, Fattizzo B. New Insights in Autoimmune Hemolytic Anemia: From Pathogenesis to Therapy Stage 1. J Clin Med. 2020 Nov 27;9(12):3859. doi: 10.3390/jcm9123859. PMID 33261023
- [Background] Kashyap R, Singh A, Kumar P. Prevalence of autoimmune hemolytic anemia in multiple myeloma: A prospective study. Asia Pac J Clin Oncol. 2016 Jun;12(2):e319-22. doi: 10.1111/ajco.12230. Epub 2014 Sep 22. PMID 25244430
- [Background] Pacca RL, Silva JBCBD, Souza KCE, Carbinatto RB. Autoimmune hemolytic anemia and hyperglobulinemia leading to the diagnosis of multiple myeloma. Rev Bras Hematol Hemoter. 2017 Oct-Dec;39(4):357-359. doi: 10.1016/j.bjhh.2017.07.005. Epub 2017 Sep 4. No abstract available. PMID 29150110
- [Background] Bird JM, Owen RG, D'Sa S, Snowden JA, Pratt G, Ashcroft J, Yong K, Cook G, Feyler S, Davies F, Morgan G, Cavenagh J, Low E, Behrens J; Haemato-oncology Task Force of British Committee for Standards in Haematology (BCSH) and UK Myeloma Forum. Guidelines for the diagnosis and management of multiple myeloma 2011. Br J Haematol. 2011 Jul;154(1):32-75. doi: 10.1111/j.1365-2141.2011.08573.x. Epub 2011 May 14. No abstract available. PMID 21569004